CLINICAL TRIAL: NCT05698602
Title: Evaluation of the Safety and Clinical Performance of NivolisMonitor and NivolisAnton: Medical Devices for Monitoring Patients Treated With Home Ventilatory Assistance Devices
Brief Title: Safety and Performance of NivolisMonitor and NivolisAnton for Monitoring Patients on Ventilatory Assistance at Home
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VIVARDIS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Nivolis
Record Dates: First submitted 2022-12-19; First posted 2023-01-26 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Insufficiency; Respiratory Failure; Home Monitoring
Keywords: Noninvasive ventilation; Nasal High Flow; Home Monitoring; Transcutaneous CO2 pressure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NivolisMonitor and NivolisAnton Arm (Experimental): For each patient enrolled in the study, a NivolisMonitor device is added to the usual ventilatory device for 3 days. NivolisMonitor is connected to the patient circuit, between the ventilatory device and the patient interface, ideally at the patient end of the circuit or possibly at the end of the breathing support device of the circuit (NIV or HDN).
  NivolisMonitor continuously measures pressure (P in cm H20) and flow (F in L.min-1) as well as temperature (T in degree Celsisus), relative humidity (RH in percent RH) and, optionally, the Fi02 (in percent).
  In addition, an overnight transcutaneous capnia recording will be performed using a Sentec SDM monitor to which a NivolisAnton device will be connected and will be able to collect data and transmit it via remote monitoring.
  Interventions: Device: NivolisMonitor; Device: NivolisAnton

INTERVENTIONS:
Device: NivolisMonitor — NivolisMonitor comprises a sensing element and controller to measure respiratory values, such as pressure and flow optionnally temperature, relative humidity and oxygen concentration, of a patient being treated with a respiratory therapy devices NIV, CPAP or HDN.
  NivolisMonitor is inserted between the respiratory assistance device and the mask or cannula inline with the standard patient circuit used routinely with the respiratory assistance device.
  NivolisMonitor functions are:
  * measure the respiratory values from the builtin sensor (Pressure, Flow, Temperature, Humidity, Oxygen fraction),
  * store the measurements in the embedded memory
  * extract from the measurement basic respiratory markers:
  * detect if and when a patient is using the respiratory assist device,
  * calculate leakage
  * calculate respiratory frequency
  * transmit the measured values via the NivolisBox component to NivolisPortal
Device: NivolisAnton — NivolisAnton device enables wireless and remote communication from tcPCO2 monitors which measure transcuteanously CO2 and O2 partial pressures in the blood (tcPCO2 & tcPO2) .
  NivolisAnton device connects to the serial port of tcPCO2 monitor, detects if the monitor is actively measuring blood gas values, collects the measurements from the monitor by following manufacturer's communication protocol and stores the collected values in its internal memory. When applicable per the manufacturer recommendations, NivolisAnton collects the values to apply the drift correction as per the manufacturer recommendations.
  NivolisAnton transmits the collected data to external receiving devices, such as Medical Devices (NivolisMonitor or another Medical Device that is granted approved data access by Vivardis) via Bluetooth or data servers (NivolisBox as an example) via WIFI. This data is thereafter transmitted by previously mentioned devices to the NivolisPortal server for archiving.

SUMMARY:
NivolisMonitor and NivolisAnton are new devices developed by Vivardis. NivolisMonitor is a generic and autonomous device for remote monitoring of ventilatory parameters generated by ventilatory assistance systems. NivolisMonitor uses its sensors to measure ventilation parameters such as pressure, flow, temperature and relative humidity, Fi02 provided by respiratory treatment devices (NIV, HDN (High Nasal Flow) and Oxygen therapy). NivolisMonitor records this data, stores it and transmits it to the healthcare professionals in charge of the patient. NivolisAnton is a medical device for telemonitoring of transcutaneous capnia, it thus helps to make recordings at the patient's home and to transmit data to healthcare professionals.

The main objective of this study is to show that the use of NivolisMonitor and NivolisAnton is done in complete safety and that the clinical performances of these two devices are achieved. For this, the data measured by NivolisMonitor will be compared with the data provided by the treatment devices used by patients at home and the data provided by NivolisAnton will be compared with the data reported by the transcutaneous capnia monitor.

The secondary objectives concern the evaluation of the acceptability/usability of the devices by patients and healthcare professionals.

This evaluation will take the form of an observational clinical study on 10 patients, including :

* a selection of patients already treated with NIV or HDN according to the inclusion/non-inclusion criteria and submission of the information note
* an inclusion visit taking place during a routine pulmonological follow-up visit for these patients with collection of the free and informed consent of each patient. The blood gas data collected during this routine consultation will be compiled in the study observation book.
* a 3-day monitoring period:

  * use over 3 days of the NivolisMonitor device at home, with on the last day the completion of the patient acceptability/usability questionnaire
  * overnight use of NivolisAnton
* a teleconsultation to close the study for each patient
* completion of the healthcare professional acceptability/usability questionnaire at the end of the study

DETAILED DESCRIPTION:
Rationale :

Since the early 2000s, there has been growing interest in remote monitoring and telemonitoring of patients with chronic respiratory pathologies, in particular patients treated with Non-Invasive Ventilation (NIV). Thus, many studies have focused on the benefits of remote monitoring or telemonitoring. Although the concept of remote home ventilation monitoring seems intuitively useful, analysis of the literature indicates a need for trials with solid evidence. In the same way, nocturnal recording of transcutaneous capnia has shown its reliability and its interest for the follow-up of patients under respiratory assistance at home.

NivolisMonitor and NivolisAnton are new devices developed by Vivardis.

Study Design :

10 patients must be included in this one arm interventional study.

Nivolis study consists in :

* a pre-inclusion visit : V0
* an inclusion visit : V1
* the 3-days study period
* a end of study visit : V2

Pre-inclusion visit V0 :

The patients included in this study are patients already treated with a Home Ventilatory Assistance (NIV) or Home Nasal High Flow device (HDN). Their care is provided by a Home Health Provider (HHP).

Pre-inclusion of patients is carried out by the investigating pulmonologist and the HHP, it aims to:

1. Check the inclusion and non-inclusion criteria
2. And if the patient is eligible, inform the patient of the study, provide him with the information note and the form for obtaining his free and informed consent.

After having been informed, the patients have a period of reflection (1 week) before the inclusion visit during which the pulmonologist will collect the free, informed and written consent of the participant.

Inclusion Visit V1 :

This visit is a classic pulmonological consultation for the follow-up of a patient with Chronic Respiratory Failure by a pulmonologist.

This visit will take place as follows:

1. Collection of the patient's free and informed consent. A copy of the information note and the signed consent is given to the participant. The original copy is kept by the investigating doctor, a third copy is kept by the sponsor.
2. The patient will benefit from his usual consultation by the pulmonologist
3. NIV or HDN device settings: NIV or HDN settings

Data collected:

* Arterial gasometry
* NIV Settings
* HDN settings
* Oxygen therapy

  3-days study period : For each patient enrolled in the study, at home, a NivolisMonitor recording for 3 days and a NivolisAnton recording for one night are performed.

The installation of NivolisMonitor and NivolisAnton is carried out by the Home Health Provider who supports the patient as part of the provision of his Ventilatory Assistance or Nasal High Flow device.

End of Study Visit V2 :

This visit is a pneumological teleconsultation for the follow-up of a patient with Respiratory sufficiency Chronic by a pulmonologist.

Data collected during this visit :

* NIV settings and usage
* HDN settings
* Sentec SDM Monitor data
* NivolisMonitor data
* NivolisAnton data
* Usability/Acceptability:

Data Management :

All data concerning visits V0, V 1, V2 will be entered into a CRF. Neither the CRF nor the database contains the identity of the patient (surname, first name). The patient is identified in these 2 documents by a number. The match between names and identification numbers is kept in another file, kept separate from medical information; He ensures the follow-up of the patients participating in the study.

The database is centralized, backed up daily. All these operations are performed continuously, that is, as the data is collected.

Statistics :

Statistical analysis of the data will be performed using IBM SPSS statistical analysis software.

All data are expressed as a mean ± standard deviation, median, frequency or percentage, if applicable.

The materiality level (level α ) is set at 0.05.

Statistical analysis includes:

* A description of patients includes:

  1. Number of patients
  2. Age, sex, weight, height, BMI
  3. Pathologies
* A description of deviations from the protocol: number and % of patients incorrectly included, patients lost at follow-up, patients who did not use the telemedicine system
* A description of all data collected during V1 and V2, as well as during the 3-day collection period.

The frequency distributions will be analyzed with the Chi² test.

For NivolisMonitor:

The Anova analysis will be used to analyze all quantitative data collected during V1 and V2 and during the 3-day collection period.

Data collected from VNI software and NivolisMonitor will be analyzed with a single-factor Anova analysis. A linear regression analysis will be conducted, in addition, a visual analysis by the Bland and Altman method will be performed.

For NivolisAnton:

The comparison between the data collected by NivolisAnton and the Sentec SDM Transcutaneous Capnia Monitor will be performed using Anova Analysis (repeated measurements), one-factor regression analysis, and Bland and Altman visual evaluation.

For the evaluation of Usability/Acceptability, the data collected and the responses to the questionnaires will be expressed in frequency (percentage).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with home ventilatory devices: NIV (Philipps Dreamstation or Resmed Lumis) or HDN

  * COPD patient treated with NIV or HDN according to current recommendations
  * Patient with Obesity Hypoventilation Syndrome treated with NIV or HDN according to current recommendations

Exclusion Criteria:

* Progressive and life-threatening condition in the short term (1 year) (cancer, rapidly progressing neuromuscular disease) (at physician's discretion)
* Patients treated with NIV other than Philipps Dreamstation or Resmed Lumis
* Hospitalization leading to NIV discontinuation for at least 1 week during the screening phase
* Person deprived of liberty
* Adult protected by law
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventilatory frequency expressed in breaths.min-1 | At the end of the 3-day monitoring period
  The values of ventilatory frequency assessed by NivolisMonitor will be compared to ventilatory frequency values measured by Resmed NIV or Philipps NIV.
  Ventilatory frequency is expressed as a median or average value, and compared according to the used NIV, respectively : Median for Resmed NIV and Average for VNI Philipps.
Leaks expressed in L.min-1 | At the end of the 3-day monitoring period
  The values of Leaks assessed by NivolisMonitor will be compared to leaks values measured by Resmed NIV or Philipps NIV.
  Leaks are expressed as a median or average value, and compared according to the used NIV, respectively : Median for Resmed NIV and Average for VNI Philipps.
Use of the device expressed in Hours | At the end of the 3-day monitoring period
  The values of Use of the NIV device assessed by NivolisMonitor will be compared to Use of the device values measured by Resmed NIV or Philipps NIV.
  Use of the device is expressed as a median or average value, and compared according to the used NIV, respectively : Median for Resmed NIV and Average for VNI Philipps.
Air Flow expressed in L.min-1 | At the end of the 3-day monitoring period
  The values of Air Flow assessed by NivolisMonitor will be compared to Air Flow values prescribed for Resmed NIV or Philipps NIV or HDN devices.
  Air Flow is expressed as a median value.
FiO2 expressed as percent | At the end of the 3-day monitoring period
  NivolisMonitor measures FiO2 values of air delivered for Resmed NIV or Philipps NIV or HDN use.
  FiO2 is expressed as a median value.
Temperature Expressed in degree Celsius | At the end of the 3-day monitoring period
  NivolisMonitor measures Temperature values of air delivered for Resmed NIV or Philipps NIV or HDN use.
  Temperature is expressed as a median value.
  Median Temperature Expressed in degree Celsius
Relative Humidity expressed as percent RH | At the end of the 3-day monitoring period
  NivolisMonitor measures relative humidity values of air delivered for Resmed NIV or Philipps NIV or HDN use.
  Relative humidity is expressed as a median value.
Device Use expressed in Hours | At the end of the 3-day monitoring period
  NivolisMonitor measures use of device values for Resmed NIV or Philipps NIV or HDN devices.
  Use of device is expressed as a median value.
TcPCO2 values expressed in mm Hg | At the end of the 3-day monitoring period
  NivolisAnton collects tcPCO2 values from Sentec SDM monitor. tcPCO2 value, collected by NivolisAnton, expressed in average during the overnight recording will be compared to tcPCO2 value measured by Sentec SDM monitor

SECONDARY OUTCOMES:
Patient Usability of NivolisMonitor | At the end of the 3-day monitoring period
  NivolisMonitor patient usability will be assessed with a usability questionnaire.
  Usability questionnaire consits in 5 questions. For each question, 6 answers are proposed ranging from Totally Agree to Totally Disagree.
Health Practitioner Usability of NivolisMonitor | At the end of the 3-day monitoring period
  NivolisMonitor health practitioner usability will be assessed with a usability questionnaire Usability questionnaire consits in 10 questions. For each question, 3 answers are proposed ranging from Completely Disagree to Totally Agree.
Health Practitioner Usability of NivolisAnton | At the end of the 3-day monitoring period
  NivolisAnton health practitioner usability will be assessed with a usability questionnaire Usability questionnaire consits in 10 questions. For each question, 3 answers are proposed ranging from Completely Disagree to Totally Agree.
tcPCO2 corrected values expressed in mm Hg | At the end of the 3-day monitoring period
  NivolisAnton collects tcPCO2 values from Sentec SDM monitor. During a night of recording with Sentec SDM monitor, a drift appears in tcPCO2 values, this drift is corrected according to a corrector factor calculated by Sentec SDM monitor at the end of the recording.
  tcPCO2 corrected value, measured by NivolisAnton, expressed in average during the overnight recording will be compared to tcPCO2 corrected value measured by Sentec SDM monitor
SaO2 expressed in % | At the end of the 3-day monitoring period
  NivolisAnton collects SaO2 values from Sentec SDM monitor. SaO2 value, collected by NivolisAnton, expressed in average during the overnight recording will be compared to SaO2 value measured by Sentec SDM monitor
  NivolisAnton : Physiological data collected during registration:
  * Arterial saturation with O 2 (SaO2) in %
  * Heart Rate (HR) in Beats Per Minute
Heart Rate (HR) in Beats Per Minute | At the end of the 3-day monitoring period
  NivolisAnton collects Heart Rate values from Sentec SDM monitor. HR value, collected by NivolisAnton, expressed in average during the overnight recording will be compared to HR value measured by Sentec SDM monitor

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, Professor, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No